CLINICAL TRIAL: NCT00354302
Title: The Influence of Five Years of Adjuvant Anastrozole or Exemestane on Bone Mineral Density In Postmenopausal Women With Primary Breast Cancer
Brief Title: Bone Mineral Density in Postmenopausal Women With Primary Breast Cancer Who Are Receiving Treatment on Clinical Trial
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: NCIC Clinical Trials Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH); North Central Cancer Treatment Group (Network); SWOG Cancer Research Network (Network)
Responsible Party: Sponsor
Organization: Canadian Cancer Trials Group (Network)
Allocation: Not Applicable | Model: Single Group | Masking: Quadruple | Purpose: Diagnostic
Other Study IDs: MA27B; CAN-NCIC-MA27B (Registry Identifier: National Cancer Institute - Physician Data Query); SWOG-NCIC-MA27B (Other: SWOG); NCCTG-NCIC-MA27B (Other: NCCTG); CAN-NCIC-BONE; CDR0000483099 (Other: PDQ)
Record Dates: First submitted 2006-07-19; First posted 2006-07-20 (Estimated); Last update posted 2020-04-02 (Actual); Status verified 2012-01

CONDITIONS: Breast Cancer; Osteoporosis
Keywords: osteoporosis; stage I breast cancer; stage II breast cancer; stage IIIA breast cancer
MeSH Terms: conditions — Breast Neoplasms; Osteoporosis | interventions — Calcium Carbonate; Calcium Citrate; Cholecalciferol; Alendronate; Calcium Gluconate; Risedronic Acid; Absorptiometry, Photon

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Dietary Supplement: calcium carbonate
Dietary Supplement: calcium citrate
Dietary Supplement: cholecalciferol
Drug: alendronate sodium
Drug: calcium gluconate
Drug: risedronate sodium
Other: laboratory biomarker analysis
Procedure: dual x-ray absorptometry

SUMMARY:
RATIONALE: Learning about the effect of exemestane and anastrozole on bone mineral density in postmenopausal women with primary breast cancer may help plan treatment, decrease the risk of broken bones, and help patients live more comfortably.

PURPOSE: This phase III trial is studying bone mineral density in postmenopausal women with primary breast cancer who are receiving treatment on clinical trial CAN-NCIC-MA27.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine whether there is a clinically relevant difference in bone mineral density (BMD) at 2 years in postmenopausal women with primary breast cancer (with or without osteopenia or osteoporosis) treated with exemestane vs anastrozole on protocol CAN-NCIC-MA27.

OUTLINE: This is a multicenter, companion study. Patients are stratified according to baseline bone mineral density (BMD) measurement (T-score* ≥ -2.0 standard deviation [SD] [no osteopenia or osteoporosis] vs T-score* < -2.0 SD).

NOTE: *The lowest of the two T-scores: L1-L4 or total hip

Blood samples for the identification of bone biomarkers (formation marker: serum amino-terminal procollagen 1 extension peptide [P1NP] and resorption marker: serum N-telopeptide) are obtained at baseline and at 6 and 12 months. BMD is determined by dual-energy x-ray absorptiometry (DEXA) at baseline and then annually for 5 years (or for as long as patient is receiving treatment on protocol CAN-NCIC-MA27).

Patients receive oral calcium and oral cholecalciferol (vitamin D) daily. Patients with osteopenia or osteoporosis (stratum II) also receive oral bisphosphonate therapy

PROJECTED ACCRUAL: A total of 408 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Enrolled in and meets eligibility requirements for protocol CAN-NCIC-MA27
* Acceptable quality dual-energy x-ray absorptiometry (DEXA) of the L1-L4 postero-anterior spine and hip within 12 weeks prior to randomization on protocol CAN-NCIC-MA27
* Hormone receptor status:

  * Estrogen receptor- and/or progesterone receptor-positive tumor

PATIENT CHARACTERISTICS:

* Female
* Postmenopausal
* No malabsorption syndrome
* No known cholecalciferol (vitamin D) deficiency, active hyper- or hypoparathyroidism, or Paget's disease
* No uncontrolled thyroid disease, Cushing's disease, or other pituitary disease
* No other bone disease (including osteomalacia or osteogenesis imperfecta)

PRIOR CONCURRENT THERAPY:

* More than 6 months since prior drugs (investigational or not), including bisphosphonates, for the prevention of osteoporosis (stratum I)
* More than 12 months since prior and no concurrent anticonvulsants
* More than 6 months since prior and no concurrent corticosteroids at doses > 5 mg/day of prednisone (or equivalent) for > 2 weeks
* More than 12 months since prior and no concurrent anabolic steroids
* No prior bisphosphonates (stratum II)
* No concurrent sodium fluoride at daily doses ≥ 5 mg/day
* No long-term (i.e., > 6 months) use of coumarins
* No concurrent drugs (investigational or not), including bisphosphonates, for the prevention of osteoporosis (for patients with no osteopenia or osteoporosis [stratum I])

Ages: 45 Years to 120 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 497 (Actual)
Dates: Start 2006-04-24 (Actual); Primary Completion 2011-03 (Actual); Study Completion 2012-01-06 (Actual)

PRIMARY OUTCOMES:
Percentage change of bone mineral density (BMD) measured at 2 years (from baseline) in the L1-L4 region of the spine and the hip | 5 years

SECONDARY OUTCOMES:
Percentage change in BMD at 5 years (from baseline) | 5 years
Mean percentage change in BMD at 1, 3, and 5 years (from baseline) | 5 years
Proportion of patients without osteopenia or osteoporosis (stratum I) who develop BMD below the absolute threshold for osteopenia (< -2.0 standard deviation below the mean), suffer any osteoporotic fracture, or have an asymptomatic fracture revealed ... | 5 years
Percentage of patients with osteopenia or osteoporosis (stratum II) who have ≥ 5% improvement of BMD at 2 years post randomization on protocol CAN-NCIC-MA27 and who have clinically apparent osteoporosis-related fracture of the long bones | 5 years
Pattern of change in bone biomarkers from baseline | 5 years
Clinical safety and tolerability of study medications | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Paul E. Goss, MD, PhD, Study Chair — Massachusetts General Hospital; James N. Ingle, MD, Study Chair — Mayo Clinic; Dawn Hershman, MD, Study Chair — Herbert Irving Comprehensive Cancer Center
Locations (13):
- Canada (13):
  - BCCA - Vancouver Cancer Centre, Vancouver, British Columbia
  - CancerCare Manitoba, Winnipeg, Manitoba
  - The Moncton Hospital, Moncton, New Brunswick
  - Atlantic Health Sciences Corporation, Saint John, New Brunswick
  - Cambridge Memorial Hospital, Cambridge, Ontario
  - Algoma District Cancer Program, Sault Ste. Marie, Ontario
  - Thunder Bay Regional Health Science Centre, Thunder Bay, Ontario
  - Odette Cancer Centre, Toronto, Ontario
  - St. Michael's Hospital, Toronto, Ontario
  - Univ. Health Network-Princess Margaret Hospital, Toronto, Ontario
  - Hopital Charles LeMoyne, Greenfield Park, Quebec
  - CHA-Hopital Du St-Sacrement, Québec, Quebec
  - Allan Blair Cancer Centre, Regina, Saskatchewan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Goss PE, Hershman DL, Cheung AM, Ingle JN, Khosla S, Stearns V, Chalchal H, Rowland K, Muss HB, Linden HM, Scher J, Pritchard KI, Elliott CR, Badovinac-Crnjevic T, St Louis J, Chapman JA, Shepherd LE. Effects of adjuvant exemestane versus anastrozole on bone mineral density for women with early breast cancer (MA.27B): a companion analysis of a randomised controlled trial. Lancet Oncol. 2014 Apr;15(4):474-82. doi: 10.1016/S1470-2045(14)70035-X. Epub 2014 Mar 11. PMID 24636210